CLINICAL TRIAL: NCT02934828
Title: A Randomized Study of Preoperative Chemotherapy or Postoperative Chemotherapy for Early Triple Negative or Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Operable Breast Cancer
Brief Title: Study of Preoperative Chemotherapy for Early Triple Negative or HER2-positive Operable Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pin Zhang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2014A04
Record Dates: First submitted 2016-08-14; First posted 2016-10-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant chemotherapy (Experimental): Neoadjuvant Chemotherapy: TNBC:paclitaxel (PTX) 175mg/m2 d1, Carboplatin area under the curve（AUC4） d2, q14d*6. HER-2 Positive BC: PTX 175mg/m2 d1, Carboplatin AUC4 d2, q14d*6, and plus Herceptin 2mg/kg qw, 6mg/kg q3w after chemotherapy until 1 year. RECIST is used once every 2 cycles. Patients will finish 6 cycles preoperative chemotherapy when CR/partial response(PR)/stable disease(SD) by RECIST without serious adverse events.
  Interventions: Drug: Neoadjuvant Chemotherapy
- postoperative chemotherapy (Active Comparator): Postoperative Chemotherapy:Standard chemotherapy regiments according to risk of recurrence: EC-P/D±H, paclitaxel and Carboplatin plus Herceptin(TCH）, EC/TC±H, and so on.
  Interventions: Drug: postoperative chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Neoadjuvant Chemotherapy: TNBC:paclitaxel (PTX) 175mg/m2 d1, Carboplatin area under the curve（AUC4） d2, q14d*6. HER-2 Positive BC: PTX 175mg/m2 d1, Carboplatin AUC4 d2, q14d*6, and plus Herceptin 2mg/kg qw, 6mg/kg q3w after chemotherapy until 1 year.
  Other Names: preoperative chemotherapy
  Arms: Neoadjuvant chemotherapy
Drug: postoperative chemotherapy — postoperative chemotherapy: EC-P/D±H, paclitaxel and Carboplatin plus Herceptin(TCH）, EC/TC±H, and so on.
  Other Names: Adjuvant Chemotherapy
  Arms: postoperative chemotherapy

SUMMARY:
The investigators research aim to explores the optimal comprehensive treatment for TNBC and her2 positive breast cancer by comparing the efficacy of neoadjuvant with that of adjuvant treatment in improvement of RFS.

DETAILED DESCRIPTION:
Neoadjuvant Chemotherapy (NCT) is a standard treatment of patients who hope breast-conserving therapy (BCT) with locally advanced inoperable breast cancer or large tumor size. it is beneficial to degrading the tumor stage, increasing the rate of surgical resection or the BCT.People who are pathological complete response (pCR) after NCT have an improvement in disease-free survival (DFS) and overall survival (OS), as well as better prognosis. Currently, breast cancer are entering into the era of molecular classification. Different molecular subtype of breast cancer showed a significant difference in prognosis; triple negative breast cancer (TNBC) and Her2 positive breast cancer are clinically relevant terms referring to a specific subtype of breast cancer with high malignant characteristics, early recurrence and metastasis, but sensitive to primary chemotherapy, proportion of which are 15% and 20% respectively. A meta analysis shows that TNBC and her2 positive breast cancer have a higher pCR than Luminal A/B, and the increasing in pCR rate means improvement in survival.

The investigators previous study indicates that paclitaxel plus carboplatin with or without trastuzumab can improve pCR and prolong RFS in TNBC and her2 positive breast cancer Comparing to adjuvant chemotherapy.

The investigators research aim to explores the optimal comprehensive treatment for TNBC and her2 positive breast cancer by comparing the efficacy of neoadjuvant with that of adjuvant treatment in improvement of RFS.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive breast cancer confirmed by pathology evaluation of core biopsy
2. Tumors must be ER/PgR status negative (immunohistochemistry（IHC） < 10%) and lack of HER2/neu overexpression or amplification as measured by local hospital pathology laboratory (IHC +/- fluorescence in situ hybridization (FISH) and IHC < 3+, and FISH < 2.2) as described in the NCCN Guidelines
3. Female between18 to 70 years of age, Eastern Cooperative Oncology Group(ECOG) Performance Status 0 or 1
4. Early-stage TNBC or HER2 positive breast cancer according to the American Joint Committee on Cancer (AJCC) Staging Manual Clinical Stage IIA or IIB, Stage IIIA operable breast cancer
5. Previously untreated
6. Adequate hematologic function (absolute neutrophil count ≥ 1,500 cells/µL; hemoglobin > 9 g/dL, platelets > 100,000/µL.)
7. Adequate hepatic function: total bilirubin ≤ upper limit of normal (ULN), serum albumin ≥≥ 3.0 g/dL, alanine aminotransferase and aspartate aminotransferase ≤ 1.5 x ULN.

Exclusion Criteria:

1. ICH:ER/PgR status positive
2. HER2 positive breast cancer Patients with reduced ejection fraction <50% are not eligible
3. Patients with second malignancies
4. Patients with bilateral breast cancer
5. allergic constitution

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) of neoadjuvant and adjuvant treatment in TNBC and her2 positive breast cancer | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pin Zhang, professor, Study Director — Chinese Academy of Medical Sciences (CAMS)
Locations (1):
- Cancer Hospital & Institute Chinese Academy of Medical Sciences (CAMS), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided